CLINICAL TRIAL: NCT04568343
Title: Evaluation of Obscure Gastrointestinal Bleeding Patients With Conventional Capsule Endoscopy and Panoramic Side View Capsule Endoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020-07-005B
Record Dates: First submitted 2020-08-06; First posted 2020-09-29 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Capsule Endoscopes
Keywords: Capsule Endoscopes
MeSH Terms: interventions — Capsule Endoscopy

STUDY DESIGN:
Intervention Model Description: The Endocapsule (EC-10) and CapsoCam Plus (Capsovision) capsule will be used. The Endocapsule is 26mm x 11mm in size and 3.3g in weight. It has 160° angle of view with 12 hours of battery life, 2 frame per second sampling rate. One antenna unit will be packed on the patient's waist during examination adjacent to a recorder. [17] The CapsoCam Plus capsule is 31mm x 11mm in size and 4g in weight. It has a field of view of 360° with at least 15 hours of battery life, takes 20 images per second maximum, (4 frames per second from each of the four cameras). No other accessories are needed during the procedure.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- small bowel bleeding patient (Experimental): with suspicious small bowel bleeding,patient will recieve Endocapsule (EC-10) and CapsoCam Plus (Capsovision) capsule later for evaluations
  Interventions: Device: Capsule endoscopy

INTERVENTIONS:
Device: Capsule endoscopy — We use two capsule endoscopy for evaluation their diagnostic yield. Patient will recieve different capsule endoscopy:The Endocapsule (EC-10) and CapsoCam Plus (Capsovision) capsule
  Other Names: The Endocapsule (EC-10) and CapsoCam Plus (Capsovision) capsule

SUMMARY:
With the development of endoscopy, patients with suspected gastrointestinal tract disease can be evaluated with further management. Upper esophageal tract including esophagus, stomach and duodenum, and colon are easily to be evaluated in daily practice. However, small bowel, located between stomach and colon, is a long tortuous organ about 4-6 meter long and causing difficulty in optical evaluation. Since Prof. Swain and Iddan invented video capsule endoscopy(VCE) from over 20 years ago.[1] VCE is increasingly used in evaluation of small bowel disease across the world.[2, 3] Originally, VCE is composed of one front lens, with flashlight and battery to take images during its passage throughout small bowel. Wireless device were also implanted for transmission of the video signal for further diagnosis.[4] In recent decades, new generation of VCE have better image quality, longer battery life and more frequent images taken. Therefore, VCE is recommended as the first line treatment in obscure gastrointestinal bleeding(OGIB) by multiple societies.[5-7] The efficacy of capsule endoscopy in evaluating patients with OGIB is good, but not perfect. The current diagnostic yield of VCE in patients with OGIB is from 35% to 77%.[8-11] Part of OGIB patients still can't be diagnosed using current conventional capsule endoscopy. The current forward looking lens may cause some difficulties, including inability to visualize the duodenal papilla, blind points missed by capsule endoscopy. In recent years, another type of panoramic side view capsule endoscopy was developed.[12] The CapsoCam Plus (Capsovision) capsule has four cameras allowing the exploration of the small bowel through 360° lateral viewing and makes papilla stably visualized. However, this system does not include a recording system so the capsule endoscope has to be collected by the patient after defecation in order for the film to be downloaded which may be a disadvantage compared with the conventional capsule endoscopy. In previous studies, the diagnostic yield of conventional capsule endoscope and panoramic side view capsule endoscope were comparable while visualization of duodenal papilla is more frequent in using panoramic side view capsule endoscopy. [13-15] However, most studies are done in single arm historical control or randomized controlled study, which may be influenced by the uneven distribution of OGIB patients in both groups. To date only one simultaneous capsule endoscopy study using both capsule endoscope in the same patient is available to data using older version of conventional capsule endoscope and panoramic side view capsule endoscope .[16] The efficiency between two capsule endoscopies were comparable in terms of diagnostic yield and image quality.

Therefore, we aimed to conduct this study to evaluate the diagnostic efficiency between two capsule endoscopies. The aim of this study was to evaluate (1) visualization of duodenal papilla (2) diagnostic concordance (kappa value) of the conventional capsule endoscopy (Olmypus endocapsule 10) and panoramic side view (CapsoCam Plus) capsule endoscopy in the same OGIB patient. The clinical experience and satisfaction of both capsule endoscope by the patient and the physicians will be also be assessed.

DETAILED DESCRIPTION:
Materials and Methods Patients 30 Patients with occult gastrointestinal bleeding aged 20-85 years old will be enrolled from Endoscopy Center for Diagnosis and Treatment, Taipei Veterans General Hospital. Patients needed to have negative esophagogastroduodenoscopy and colonoscopy for potential bleeding source within 12 months prior to the capsule examination. Patient with suspected or confirmed gastrointestinal tract obstruction, pacemaker use or unwilling to swallow the capsule endoscope will be excluded. Female at child bearing age will receive urine HCG test for pregnancy evaluation. Pregnant patients will be excluded. All patients will be given informed consent before inclusion.

Capsule Endoscopy procedure The Endocapsule (EC-10) and CapsoCam Plus (Capsovision) capsule will be used. The Endocapsule is 26mm x 11mm in size and 3.3g in weight. It has 160° angle of view with 12 hours of battery life, 2 frame per second sampling rate. One antenna unit will be packed on the patient's waist during examination adjacent to a recorder. [17] The CapsoCam Plus capsule is 31mm x 11mm in size and 4g in weight. It has a field of view of 360° with at least 15 hours of battery life, takes 20 images per second maximum, (4 frames per second from each of the four cameras). No other accessories are needed during the procedure.

Small-bowel preparation will be performed in patients before capsule ingestion as routine practice and previously published guidelines. [19] The patients will take one pack of GI-Klean powder(polyethylene glycol) in 1000ml water followed by 1000ml water at 6-8 pm the night before capsule endoscopy. Then they will take another pack of GI-Klean powder(polyethylene glycol) in 1000ml water followed by 1000ml water at 5AM on the morning on the day of capsule endoscopy.

On the day of examination, the patients will take 10ml of simethicone fluid first. Then they'll ingest the two capsules, with 1.5 hour between and in a randomized order (using sealed envelopes). After capsule endoscopy entered small bowel, the patient will take a light meal at least 4 hours after the 2nd capsule endoscope ingestion. They'll take dinner as usual. The capsule endoscope will be collected by the patient using a specified capsule collecting system during defecation. If no capsule endoscope was noted in the stool in 3 days. The patient will received through 20mg sennosides on the 3rd night. The patients will return back the capsule endoscope, antenna and recorder after getting the capsule endoscope. For patient who didn't collect capsule endoscope in 15 days, abdominal x-ray plain film will be taken to evaluate the status of capsule endoscope.

Capsule endoscopy review For each case, the two capsule films will read in a randomized order by three experienced physicians (one >250 VCE examinations, two >100 VCE examinations). None of the physicians had experience of panoramic side view capsule endoscopy(<5) before this study. The two readings will be done blindly. The reading frames will be were available to each reader, and suggested not faster than a rate of 15 images per second. The cases will be classified into concordant positive, concordant negative, and discordant cases. For discordant cases, a third reviewer will conduct the clarification of the CE images for confirmation and confirmed during a conference by all three experienced readers. An image per image comparison will be performed and the complete film will be read a second time when necessary.

The primary outcome of the study will be (1) ampulla of the vater detection rate and (2) the concordance between the two capsule examinations with a kappa value>0.5. The secondary outcomes will be the small bowel cleansing quality, technical failure rate, transit and operation time, capsule endoscopy completion rate, video record reliability, diagnostic yield, safety profile and the physicians' and patients' satisfaction with the capsule endoscopy.

The definition of the outcome measurement will be defined as following:

1. Ampulla of Vater detection rate: the number of examinations in which the ampulla was clearly identified over the number of the overall number of patients receiving VCE
2. Data interpretation: All endoscopic findings will be systemically recorded according to location, endoscopic features and clinical significance, and in relation to procedure indications, as P0 (low probability), P1 (intermediate pcccrobability), or P2 (high probability) as in previous descriptions [18]. Nonsignificant (P0) lesions and images located outside the small intestine were not considered. For per patient analysis, the final diagnosis of P1 or P2 lesions will be used according to the description of the most important or the most relevant lesion or group of lesions. The sensitivity of each capsule examination will be assessed, with true-positive cases being calculated as the sum of positive cases obtained from the Endocapsule 10 or CapsoCam plus readings, including expert review of discordant cases. In a per lesion analysis, each lesion (up to three main lesions found from capsule reading) or group of lesions will be analyzed independently.
3. Diagnostic Yield: VCE will be defined as 'positive' when at least one clinically significant finding (P2) was identified; the rate of "positive" VCE (ie, DY) will be calculated.
4. Small bowel cleansing quality: The small-bowel cleansing will be scored by estimating the amount of clearly visible mucosa using the scale proposed by Esaki et al. [19]. The images of the small intestine will equally be separated into 3 segments according to SBTT. The cleansing quality will be graded according to fluid transparency and mucosal invisibility. The fluid transparency will be graded into grade 1, Clear fluid without obscuring vision, grade 2 Slightly dark fluid minimally obscuring vision, grade 3 Opaque fluid partly obscuring vision and grade 4 Turbid fluid severely obscuring vision. The mucosal invisibility will be graded as Grade 1, <5% in duration of 50% bubbles or residues, grade 2 5%-15%, grade 3 15%-25% and grade 4 >25%. The overall image quality will be categorized into Grade A 3-5, Grade B 6-8 and Grade C 9-12.
5. Technical failure: it will be defined as any encountered technical problem due to one or more system components (such as capsule device, downloading system, and/or workstation) influencing the generation of the video.
6. Transit and operating times: Gastric transit time, will be defined as the time between the first and the last gastric image. Small-bowel transit time (SBTT), will be defined as the timeframe between the first and the last small-bowel image. Total capsule endoscope time will be defined as the time between the first and the last image captured by the capsule. Reading time will be defined as the time doctors read the full capsule endoscopic images.
7. Capsule endoscopy completion rate: the number of examinations in which the colon was reached during the operating time over the overall number of patients receiving VCE.
8. Video record reliability: the video record reliability will be evaluated according to a quantitative scoring system as described before, the images of the small intestine will equally be separated into 3 segments according to SBTT. The scoring system is defined as following: 3 points - excellent: when less than 5 total frames and no consecutive non-evaluable frames were observed. 2 points - good: when ≥5 to <10 total frames or one sequence with <5 consecutive non-evaluable frames were observed. 1 point - fair: when ≥10 to <15 total frames, or one sequence with <10 consecutive non-evaluable frames were observed. 0 points - poor: when ≥15 total frames, or multiple sequences, or one sequence with ≥10 consecutive non-evaluable frames were observed.[13] The video record reliability will be evaluated only in completed capsule endoscopy cases.
9. Safety profile: As reported in previous studies on front-viewing capsules [1,21], we will focus our attention on capsule aspiration, at time of ingestion, and capsule retention. Capsule retention will be defined as the persistence of the capsule within the patient's intestinal tract, evaluated by an abdominal x-ray plain film, 15 days after capsule ingestion. There is 1 % chance of capsule endoscope retention in gastrointestinal tract and patients in whom the capsule was retrieved by elective surgery and/or by endoscopic procedures will also be considered as capsule retention. Any other incident and/or adverse event, reported as potentially related to VCE by the local investigator, will be documented and classified according to previously published international guidelines.[20]
10. Patients' Satisfaction Questionnaire: For evaluation of the convenience and satisfaction of the patient about two capsule endoscopy, the patient will be asked to fill a questionnaire about the capsule endoscopy procedure after the capsule endoscopy procedure.
11. Physician's satisfaction evaluation: For evaluation and further recommendation of the physician on two different capsule endoscopy about their convenience and efficacy, physician will be asked to fill up a satisfaction sheet after capsule endoscopy procedure and image analysis.

3. Statistical analysis In a recent study, the detection rate of ampulla vater is 81.7 % in panoramic view capsule endoscopy and 9.6% in conventional capsule endoscopy. 18 patients are needed to give the study 80% power atα=0.05%.[21] For evaluation of interobserver agreement, the calculated sample size for detection of was 27 patients in order to obtain a satisfying estimation of concordance, with an 80% power, of the kappa interobserver agreement coefficient between paired (Endocapsule 10(Olympus) and CapsoCam Plus(Capsovision)) capsule readings, taking into account the positive diagnostic yield of VCE in OGIB reaches about 60%. With an estimation of 10% dropout rate, 30 patients will be needed for this study.

The median with inter-quartile range (IQR) and range will be provided for non-normally distributed variables, whereas the mean ± standard deviation (SD) for normally distributed variables. The paired T test will be used to compare technical outcomes among two capsule endoscopies (ie, operative time and video records reliability). The 2-tailed Fisher exact test will be used to compare the diagnostic yield. To compare the sensitivity of Endocapsule 10and CapsoCam Plus, a Mac-Nemar test will be used with the exact test of the binomial law.

For statistical analysis, SPSS software version 26.0 (SPSS Inc., Chicago, Illinois, USA) in a Windows XP (Microsoft, Seattle, Washington,USA) environment will be used. A P value of <0.05 was considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients needed to have negative esophagogastroduodenoscopy and colonoscopy for potential bleeding source within 12 months prior to the capsule examination

Exclusion Criteria:

* suspected or confirmed gastrointestinal tract obstruction, pacemaker use or unwilling to swallow the capsule endoscope

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-06-06 (Estimated); Study Completion 2022-06-06 (Estimated)

PRIMARY OUTCOMES:
Ampulla of Vater detection rate | 24 months
  rate of specificaly detect Ampulla of Vater the number of examinations in which the ampulla was clearly identified over the number of the overall number of patients receiving VCE
the concordance between the two capsule examinations with a kappa value>0.5 | 24 months
  concordance between the two capsule All endoscopic findings will be systemically recorded according to location, endoscopic features and clinical significance, and in relation to procedure indications, as P0 (low probability), P1 (intermediate pcccrobability), or P2 (high probability) as in previous descriptions [18]. Nonsignificant (P0) lesions and images located outside the small intestine were not considered. For per patient analysis, the final diagnosis of P1 or P2 lesions will be used according to the description of the most important or the most relevant lesion or group of lesions. The sensitivity of each capsule examination will be assessed, with true-positive cases being calculated as the sum of positive cases obtained from the Endocapsule 10 or CapsoCam plus readings, including expert review of discordant cases. In a per lesion analysis, each lesion (up to three main lesions found from capsule reading) or group of lesions will be analyzed independently.

SECONDARY OUTCOMES:
small bowel cleansing quality | 24 months
  The small-bowel cleansing will be scored by estimating the amount of clearly visible mucosa using the scale proposed by Esaki et al. The images of the small intestine will equally be separated into 3 segments according to SBTT. The cleansing quality will be graded according to fluid transparency and mucosal invisibility. The fluid transparency will be graded into grade 1, Clear fluid without obscuring vision, grade 2 Slightly dark fluid minimally obscuring vision, grade 3 Opaque fluid partly obscuring vision and grade 4 Turbid fluid severely obscuring vision. The mucosal invisibility will be graded as Grade 1, <5% in duration of 50% bubbles or residues, grade 2 5%-15%, grade 3 15%-25% and grade 4 >25%. The overall image quality will be categorized into Grade A 3-5, Grade B 6-8 and Grade C 9-12.
technical failure rate | 24 months
  it will be defined as any encountered technical problem due to one or more system components (such as capsule device, downloading system, and/or workstation) influencing the generation of the video.
transit and operation time | 24 months
  Gastric transit time, will be defined as the time between the first and the last gastric image. Small-bowel transit time (SBTT), will be defined as the timeframe between the first and the last small-bowel image. Total capsule endoscope time will be defined as the time between the first and the last image captured by the capsule. Reading time will be defined as the time doctors read the full capsule endoscopic images.
capsule endoscopy completion rate | 24 months
  the number of examinations in which the colon was reached during the operating time over the overall number of patients receiving VCE.
video record reliability | 24 months
  the video record reliability will be evaluated according to a quantitative scoring system as described before, the images of the small intestine will equally be separated into 3 segments according to SBTT. The scoring system is defined as following: 3 points - excellent: when less than 5 total frames and no consecutive non-evaluable frames were observed. 2 points - good: when ≥5 to <10 total frames or one sequence with <5 consecutive non-evaluable frames were observed. 1 point - fair: when ≥10 to <15 total frames, or one sequence with <10 consecutive non-evaluable frames were observed. 0 points - poor: when ≥15 total frames, or multiple sequences, or one sequence with ≥10 consecutive non-evaluable frames were observed. The video record reliability will be evaluated only in completed capsule endoscopy cases.
diagnostic yield | 24 months
  VCE will be defined as 'positive' when at least one clinically significant finding (P2) was identified; the rate of "positive" VCE (ie, DY) will be calculated.
the physicians' and patients' satisfaction with the capsule endoscopy | 24 months
  For evaluation of the convenience and satisfaction of the patient and physicians about two capsule endoscopy, the physician and patient will be asked to fill a questionnaire about the capsule endoscopy procedure after the capsule endoscopy procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Gastroenterology, Department of Medicine, Taipei Veterans General Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Iddan G, Meron G, Glukhovsky A, Swain P. Wireless capsule endoscopy. Nature. 2000 May 25;405(6785):417. doi: 10.1038/35013140. No abstract available. PMID 10839527
- [Background] Rondonotti E, Spada C, Adler S, May A, Despott EJ, Koulaouzidis A, Panter S, Domagk D, Fernandez-Urien I, Rahmi G, Riccioni ME, van Hooft JE, Hassan C, Pennazio M. Small-bowel capsule endoscopy and device-assisted enteroscopy for diagnosis and treatment of small-bowel disorders: European Society of Gastrointestinal Endoscopy (ESGE) Technical Review. Endoscopy. 2018 Apr;50(4):423-446. doi: 10.1055/a-0576-0566. Epub 2018 Mar 14. PMID 29539652
- [Background] Enns RA, Hookey L, Armstrong D, Bernstein CN, Heitman SJ, Teshima C, Leontiadis GI, Tse F, Sadowski D. Clinical Practice Guidelines for the Use of Video Capsule Endoscopy. Gastroenterology. 2017 Feb;152(3):497-514. doi: 10.1053/j.gastro.2016.12.032. Epub 2017 Jan 4. PMID 28063287
- [Background] Singeap AM, Stanciu C, Trifan A. Capsule endoscopy: The road ahead. World J Gastroenterol. 2016 Jan 7;22(1):369-78. doi: 10.3748/wjg.v22.i1.369. PMID 26755883
- [Background] ASGE Standards of Practice Committee; Gurudu SR, Bruining DH, Acosta RD, Eloubeidi MA, Faulx AL, Khashab MA, Kothari S, Lightdale JR, Muthusamy VR, Yang J, DeWitt JM. The role of endoscopy in the management of suspected small-bowel bleeding. Gastrointest Endosc. 2017 Jan;85(1):22-31. doi: 10.1016/j.gie.2016.06.013. Epub 2016 Jun 30. No abstract available. PMID 27374798
- [Background] Pennazio M, Spada C, Eliakim R, Keuchel M, May A, Mulder CJ, Rondonotti E, Adler SN, Albert J, Baltes P, Barbaro F, Cellier C, Charton JP, Delvaux M, Despott EJ, Domagk D, Klein A, McAlindon M, Rosa B, Rowse G, Sanders DS, Saurin JC, Sidhu R, Dumonceau JM, Hassan C, Gralnek IM. Small-bowel capsule endoscopy and device-assisted enteroscopy for diagnosis and treatment of small-bowel disorders: European Society of Gastrointestinal Endoscopy (ESGE) Clinical Guideline. Endoscopy. 2015 Apr;47(4):352-76. doi: 10.1055/s-0034-1391855. Epub 2015 Mar 31. PMID 25826168
- [Background] Gerson LB, Fidler JL, Cave DR, Leighton JA. ACG Clinical Guideline: Diagnosis and Management of Small Bowel Bleeding. Am J Gastroenterol. 2015 Sep;110(9):1265-87; quiz 1288. doi: 10.1038/ajg.2015.246. Epub 2015 Aug 25. PMID 26303132
- [Background] Lecleire S, Iwanicki-Caron I, Di-Fiore A, Elie C, Alhameedi R, Ramirez S, Herve S, Ben-Soussan E, Ducrotte P, Antonietti M. Yield and impact of emergency capsule enteroscopy in severe obscure-overt gastrointestinal bleeding. Endoscopy. 2012 Apr;44(4):337-42. doi: 10.1055/s-0031-1291614. Epub 2012 Mar 2. PMID 22389234
- [Background] Estevez E, Gonzalez-Conde B, Vazquez-Iglesias JL, de Los Angeles Vazquez-Millan M, Pertega S, Alonso PA, Clofent J, Santos E, Ulla JL, Sanchez E. Diagnostic yield and clinical outcomes after capsule endoscopy in 100 consecutive patients with obscure gastrointestinal bleeding. Eur J Gastroenterol Hepatol. 2006 Aug;18(8):881-8. doi: 10.1097/00042737-200608000-00014. PMID 16825907
- [Background] Robinson CA, Jackson C, Condon D, Gerson LB. Impact of inpatient status and gender on small-bowel capsule endoscopy findings. Gastrointest Endosc. 2011 Nov;74(5):1061-6. doi: 10.1016/j.gie.2011.07.019. Epub 2011 Sep 15. PMID 21924720
- [Background] Albert JG, Schulbe R, Hahn L, Heinig D, Schoppmeyer K, Porst H, Lorenz R, Plauth M, Dollinger MM, Mossner J, Caca K, Fleig WE. Impact of capsule endoscopy on outcome in mid-intestinal bleeding: a multicentre cohort study in 285 patients. Eur J Gastroenterol Hepatol. 2008 Oct;20(10):971-7. doi: 10.1097/MEG.0b013e3282fb2a53. PMID 18787463
- [Background] Friedrich K, Gehrke S, Stremmel W, Sieg A. First clinical trial of a newly developed capsule endoscope with panoramic side view for small bowel: a pilot study. J Gastroenterol Hepatol. 2013 Sep;28(9):1496-501. doi: 10.1111/jgh.12280. PMID 23701674
- [Background] Tontini GE, Wiedbrauck F, Cavallaro F, Koulaouzidis A, Marino R, Pastorelli L, Spina L, McAlindon ME, Leoni P, Vitagliano P, Cadoni S, Rondonotti E, Vecchi M. Small-bowel capsule endoscopy with panoramic view: results of the first multicenter, observational study (with videos). Gastrointest Endosc. 2017 Feb;85(2):401-408.e2. doi: 10.1016/j.gie.2016.07.063. Epub 2016 Aug 8. PMID 27515129
- [Background] Branchi F, Ferretti F, Orlando S, Tontini GE, Penagini R, Vecchi M, Elli L. Small-bowel capsule endoscopy in patients with celiac disease, axial versus lateral/panoramic view: Results from a prospective randomized trial. Dig Endosc. 2020 Jul;32(5):778-784. doi: 10.1111/den.13575. Epub 2019 Nov 26. PMID 31680344
- [Background] Zwinger LL, Siegmund B, Stroux A, Adler A, Veltzke-Schlieker W, Wentrup R, Jurgensen C, Wiedenmann B, Wiedbrauck F, Hollerbach S, Liceni T, Bojarski C. CapsoCam SV-1 Versus PillCam SB 3 in the Detection of Obscure Gastrointestinal Bleeding: Results of a Prospective Randomized Comparative Multicenter Study. J Clin Gastroenterol. 2019 Mar;53(3):e101-e106. doi: 10.1097/MCG.0000000000000994. PMID 29369240
- [Background] Pioche M, Vanbiervliet G, Jacob P, Duburque C, Gincul R, Filoche B, Daudet J, Filippi J, Saurin JC; French Society of Digestive Endoscopy (SFED). Prospective randomized comparison between axial- and lateral-viewing capsule endoscopy systems in patients with obscure digestive bleeding. Endoscopy. 2014 Jun;46(6):479-84. doi: 10.1055/s-0033-1358832. Epub 2013 Nov 27. PMID 24285122
- [Background] Hosoe N, Watanabe K, Miyazaki T, Shimatani M, Wakamatsu T, Okazaki K, Esaki M, Matsumoto T, Abe T, Kanai T, Ohtsuka K, Watanabe M, Ikeda K, Tajiri H, Ohmiya N, Nakamura M, Goto H, Tsujikawa T, Ogata H. Evaluation of performance of the Omni mode for detecting video capsule endoscopy images: A multicenter randomized controlled trial. Endosc Int Open. 2016 Aug;4(8):E878-82. doi: 10.1055/s-0042-111389. Epub 2016 Aug 8. PMID 27540577
- [Background] Saurin JC, Delvaux M, Gaudin JL, Fassler I, Villarejo J, Vahedi K, Bitoun A, Canard JM, Souquet JC, Ponchon T, Florent C, Gay G. Diagnostic value of endoscopic capsule in patients with obscure digestive bleeding: blinded comparison with video push-enteroscopy. Endoscopy. 2003 Jul;35(7):576-84. doi: 10.1055/s-2003-40244. PMID 12822092
- [Background] Esaki M, Matsumoto T, Kudo T, Yanaru-Fujisawa R, Nakamura S, Iida M. Bowel preparations for capsule endoscopy: a comparison between simethicone and magnesium citrate. Gastrointest Endosc. 2009 Jan;69(1):94-101. doi: 10.1016/j.gie.2008.04.054. Epub 2008 Aug 16. PMID 18710720
- [Background] Spada C, McNamara D, Despott EJ, Adler S, Cash BD, Fernandez-Urien I, Ivekovic H, Keuchel M, McAlindon M, Saurin JC, Panter S, Bellisario C, Minozzi S, Senore C, Bennett C, Bretthauer M, Dinis-Ribeiro M, Domagk D, Hassan C, Kaminski MF, Rees CJ, Valori R, Bisschops R, Rutter MD. Performance measures for small-bowel endoscopy: a European Society of Gastrointestinal Endoscopy (ESGE) Quality Improvement Initiative. Endoscopy. 2019 Jun;51(6):574-598. doi: 10.1055/a-0889-9586. Epub 2019 May 10. PMID 31075800
- [Background] Pachofszky T., H.P., Madl C., World's largest series with CapsoCam®. Feasibility, completion and detection rate of the new Generation of capsule endoscope with a 360° lateral panoramic view - A single center retrospective study., in UEG Week. 2019: Barcelona, Spain